CLINICAL TRIAL: NCT00511394
Title: Acute Hemodynamic Effects of Albumin Versus Normal Saline in Patients With Cirrhosis With Ascites: A Randomized Controlled Trial
Brief Title: Acute Hemodynamics of Albumin Versus Normal Saline in Cirrhosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Dr S K Sarin, G B Pant Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2007-PHT-01
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Cirrhosis; Ascites
Keywords: Decompensated Cirrhosis with Ascites
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Serum Albumin, Human; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): Infusion of 100 mL of 20% Albumin
  Interventions: Drug: 20% Human Albumin
- II (Placebo Comparator): 100 mL Normal Saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: 20% Human Albumin — Infusion of 100 mL of 20% Albumin over 3 hours
  Arms: I
Drug: Normal Saline — Infusion of 100 mL of Normal Saline
  Arms: II

SUMMARY:
Cirrhosis is frequently complicated by derangement of body fluid homeostasis resulting in accumulation of large amounts of extracellular fluid in the peritoneal cavity (ascites) and interstitial tissue (edema). Studies showed that patients with cirrhosis and ascites have marked circulatory dysfunction. Albumin infusions have been used for many years in the management of patients with cirrhosis and ascites in an attempt to reduce the formation of ascites and/or improve circulatory and renal function. While some of these indications for albumin infusions are supported by the results of randomised studies, others are based on clinical experience and have not been proved in prospective investigations. Therefore, the use of albumin infusions in patients with cirrhosis is controversial. Recently, this debate has been fostered by the high cost and limited availability of albumin and the results of a meta-analysis showing that albumin administration may increase mortality in critically ill patients. In cirrhotics, there is a significant improvement in the low effective arterial blood volume, which may be important in the prevention of circulatory dysfunction and in preventing renal impairment. However, in an already fluid overload state such as that of cirrhosis, albumin infusion predisposes the individual to develop pulmonary edema. There is no study demonstrating acute effect of albumin infusion on hemodynamic parameters, in cirrhotic patients. Neither is there is data concerning comparison between albumin and normal saline. It is postulated that it may increase portal pressure thereby increasing the risk of variceal bleed. This study hypothesizes that albumin infusion might lead to alteration in portal and pulmonary hemodynamics in decompensated cirrhotic patients. Included patients of cirrhosis with ascites (based on inclusion and exclusion criteria) will undergo baseline investigations (systemic hemodynamics, pulmonary hemodynamics, portal hemodynamics). They will be randomized into two groups, each of 8. One group will receive infusion of 100 ml 20% albumin over 3 hours, and the other will receive infusion of 100 ml normal saline over 3 hours. Repeat hemodynamic studies will be performed after the infusion finishes. All results will be expressed as mean ± SD or frequency (%). Comparisons will be performed by the Student's t test or with the Wilcoxon's test

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cirrhosis with ascites admitted to the GE ward
2. They require intravenous albumin therapy, for the management of their cirrhotic ascites
3. Their serum albumin <2.8 g/dL

Exclusion Criteria:

1. Cirrhotics without ascites
2. Acute on chronic liver failure
3. Serum bilirubin >3 mg/dL
4. Hepatorenal syndrome
5. Patients suffering from heart disease, history of allergy to albumin, pregnant women, hypertension, chronic nephritis
6. Lack of informed written consent

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Immediate change in mean arterial pressure, cardiac output, systemic vascular resistance, pulmonary capillary wedge pressure, pulmonary vascular resistance and HVPG on infusion of 100 ml of 20% albumin or normal saline in decompensated cirrhotics | Immediately after 3 hours of infusion

SECONDARY OUTCOMES:
Adverse effects to the drug (albumin or normal saline) | During or immediately after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD, DM, Principal Investigator — Govind Ballabh Pant Hospital
Locations (1):
- Department of Gastroenterology, G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India